CLINICAL TRIAL: NCT05324163
Title: A Phase 3, Multicenter, Double-blind and Placebo and Active Control Study to Evaluate the Efficacy and Safety of X0002 Spray in Treatment of Subjects With Osteoarthritis of the Knee
Brief Title: Evaluate Efficacy and Safety of X0002 in Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu XinChen-Techfields Pharma Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TFR-X0002-301
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2022-05

CONDITIONS: KNEE OSTEOARTHRITIS
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Drug Evaluation; Celecoxib

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- X0002 spray group (Experimental): X0002 spray 17.5mg, twice a day; Celecoxib placebo 200mg, once a day
  Interventions: Drug: X0002 Spray; Drug: placebo
- Celecoxib capsule Group: (Active Comparator): X0002 spray placebo 17.5 mg, twice a day; Celecoxib capsule 200mg, once a day
  Interventions: Drug: Celecoxib capsules; Drug: placebo
- The placebo group (Placebo Comparator): X0002 spray placebo 17.5 mg, twice a day; Celecoxib placebo 200mg, once a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: X0002 Spray — X0002 spray 17.5mg, twice a day; Celecoxib placebo 200mg, once a day
  Other Names: Test drug
  Arms: X0002 spray group
Drug: Celecoxib capsules — X0002 spray placebo 17.5 mg, twice a day; Celecoxib capsule 200mg, once a day
  Other Names: Active comparator
  Arms: Celecoxib capsule Group:
Drug: placebo — X0002 spray placebo 17.5 mg, twice a day; Celecoxibplacebo 200mg, once a day
  Other Names: Placebo Spray

SUMMARY:
This study is a randomized, double-blind clinical trial in a Chinese population

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-positive, phase iii study evaluating the efficacy and safety of brothamine hydrochloride spray in patients with knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria before entering the study:

  1. Aged between 40 and 75 years old.
  2. A diagnosis of primary knee joint must be made by clinical and/or radiographic examination according to American College of Rheumatology standards

     Osteoarthritis (OA), meeting at least 4 of the following 6 criteria:

     ● Age ≥50

     Solution Number: TFR-X0002-301 Version 1.0 Date 2021-06-07

  * Rigidity lasting less than 30 minutes after waking up in the morning
  * (joint) twist pronunciation
  * There is bone tenderness
  * Bony enlargement
  * No joint heating

    3. The history of clinical symptoms of OA of knee joint should be ≥6 months, and X-ray film of knee joint can be provided to confirm the presence of bone

Hyperplasia or degeneration.

4. Knee pain during standing, walking, and/or sports for at least 14 days in the 1 month prior to screening

Pain.

5. During the 7 days prior to randomization, knee pain was not treated with analgesics (study designated salvage)

Excluding drugs), VAS score of 100mm, ≥40mm and ≤90mm for at least 5 days (as recorded on the subject's diary card).

6. At baseline visit (day 1), the mean WOMAC pain score for the target knee must be ≥40mm and ≤90mm.

7. Women in the study had to be infertile (defined as at least 1 year after menopause or having been sterilized)

Lateral tubal ligation, bilateral oophorectomy, or total hysterectomy]), or willing to perform the following

1 less medically acceptable method of birth control: ● Use hormonal contraceptive methods, such as oral, implanted, injected, vaginal ring,

Or percutaneous use of medical contraception for at least 1 full cycle (based on the subject's usual menstrual cycle).

* Intrauterine device.
* Two-barrier method (condom, sponge, or diaphragm with spermicide gel/cream).

  8. Subjects will avoid non-habituation from the first visit during the screening period through the entire study treatment period

Physical activity (e.g., starting a new weight lifting exercise).

9. Subjects were in good health except knee OA.

10. Subject is able to provide written signed and dated informed consent.

11. Be able to understand and be willing to fully comply with research process and protocol requirements.

Exclusion Criteria:

* 1. Pelecoxib, any other NSaids, aspirin, acetaminophen, sulfa drugs

Or the presence or history of alcohol allergy; Subjects are intolerant to or have used NSAIDs regularly

NSAIDs drugs treat OA, but the effect is not good.

2. Subject has a history of chronic pain (e.g., rheumatoid arthritis, psoriatic arthritis, gout joints)

Inflammation, fibromyalgia), or other conditions that may affect the target knee function and pain assessment (e.g., bone

Necrosis, cartilage calcification).

3. Subjects' knee joints were secondary OA, or OA of lower limb joints other than knee joints, according to the investigator

Judgment may affect the assessment of knee pain and function.

4. Have a history of knee replacement, arthroplasty or other knee surgery.

5. As determined by the investigator, subjects had significant injury involving the target knee in the 6 months prior to screening.

6. Subjects' knee joint on or near the knee during the screening period or before the first use of the investigational drug (day 1)

Skin lesions or cuts.

7. Subjects had used opioids or glucocorticoid stimulation for the target knee in the 30 days prior to screening

Element; Or requiring long-term treatment with opioids or glucocorticoids during the study period.

8. Subjects received intraknee injections of steroids, hyaluronic acid, or adhesives within 3 months prior to screening

(e.g., Cinvicol ®).

9. Subjects had asthma and required systemic glucocorticoid therapy (only with inhaled glucocorticoid therapy)

Asthma patients are eligible).

10. Subjects 1 month prior to screening, except for aspirin not exceeding 325 mg/ day for heart disease prevention

He was given antithrombotic drugs.

11. Subjects had active peptic ulcer in the 6 months prior to screening or gastrointestinal tract in the 5 years prior to screening

A history of blood.

12. Subject is receiving systemic chemotherapy for any type of active malignancy; Or 5 years prior to screening

Within, cancer was diagnosed (but not squamous cell carcinoma or basal cell carcinoma of the skin).

13. Subject will, in the investigator's judgment, have any clinically significant cardiac, respiratory, or mental instability

Diseases of the menstrual, immunological, blood, or kidney, or other physical, medical, ecg, or laboratory tests

Abnormalities of clinical significance that affect the evaluation of safety and efficacy. Defined as:

● Detection value of aspartate aminotransferase, alanine aminotransferase and lactate dehydrogenase ≥3× upper limit of normal value [ULN]; ● Creatinine or total bilirubin ≥1.5 × ULN; ● Hemoglobin < 10g/dL; ● Screening visit, or baseline visit (day 1). Fecal occult blood test is positive; ● Ecg abnormalities with clinical significance, including but not limited to QTc interphase abnormalities (QTc prolongidine)

Meaning male or female > 480 ms);

● uncontrolled hypertension was defined as systolic blood pressure > 170mmHg or diastolic blood pressure > 105 mmHg.

14. Subjects known to abuse alcohol or other drugs.

15. Subjects have participated in a clinical trial for brothamine hydrochloride spray or have participated in any of the trials within 1 month prior to screening

Other clinical trials, or screening fashionable drugs in other clinical trials within the 5 metabolic half-lives.

16. Female subjects, who are pregnant, planning to be pregnant, or breastfeeding.

17. The subject has an employee or immediate family relationship with the investigator.

18. Subject is unable to make or receive phone calls and/or is technically unavailable.

19. The investigator considered that the subject had conditions that were inappropriate for clinical trial participation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of ibuprofen hydrochloride spray in the treatment of subjects' target knee osteoarthritis when compared with celecoxib capsules at 12 weeks of treatment with ibuprofen hydrochloride spray. | week 12
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.

SECONDARY OUTCOMES:
Changes in WOMAC pain Scale scores for OA of the target knee compared to baseline at 1, 2, 4, and 8 weeks of treatment | week1、week2、week4、week8
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
At 1, 2, 4, 8, and 12 weeks of treatment, changes in the WOMAC Rigidity Scale score for OA of the target knee compared to baseline | week1、week2、week4、week8
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
Changes in WOMAC Daily Activity Scale scores for target knee OA compared to baseline at weeks 1, 2, 4, 8, and 12 of treatment | week1、week2、week4、week8
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
Changes in total WOMAC score for knee OA at 1, 2, 4, 8, and 12 weeks of treatment compared to baseline | week1、week2、week4、week8
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
At 1, 2, 4, 8, and 12 weeks of treatment, subjects self-assessed changes in OA of the target knee compared to baseline | week1、week2、week4、week8
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
At 1, 2, 4, 8, and 12 weeks of treatment, subjects themselves assessed the response of target knee OA to treatment (compared to baseline) | week1、week2、week4、week8
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
Changes in daily doses of salvage analgesics (acetaminophen) compared to baseline at 1, 2, 4, 8, and 12 weeks of treatment | week1、week2、week4、week8
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.

OTHER OUTCOMES:
Change in the WOMAC pain Scale score of the subject's target knee OA from baseline at week 14 (or 2 weeks after the last medication) | week14
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
At 15min, 30min, 1h and 3h after the first, second and third days of treatment, the VAS score of OA of the target knee joint was changed from baseline | 15min, 30min, 1h and 3h after the first, second and third days of treatment
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.
Changes in subjects' joint cavity effusion at week 12 compared to baseline (only for some subjects) | weer12
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) has been used to assess subjects with OA of the hip or knee and consists of 24 questions in subscales measuring 3 concepts: pain, stiffness, and physical function. These questions measure the amount of pain, degree of difficulty in completing various day-to-day activities, and stiffness experienced in the hip or knee. Usually subject self-administered. A single question has 100 grades, where 0 = very good and 100 = very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: xiaofeng zeng, Principal Investigator — Study Principal Investigator
Locations (1):
- China,Beijing, Beijing, China

IPD SHARING:
Plan to Share IPD: No